CLINICAL TRIAL: NCT00413517
Title: Evaluation of Epi-lasik in U.S. Army Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WRAMC WU # 06-23020
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: Myopia
Keywords: Naturally occurring myopia with or without astigmatism
MeSH Terms: conditions — Myopia

INTERVENTIONS:
Procedure: Epi-Lasik — A vision correcting surgery

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Epi-Lasik in U.S. Army personnel who have naturally occurring myopia with or without astigmatism. The data from this control group will be collected in such a way as to be comparable to data sets from study groups undergoing wavefront guided PRK, conventional PRK, and related laser refractive surgery procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Active duty US Army Soldiers eligible for care at WRAMC
2. Male or female, of any race, and at least 21 years old at the time of the pre-operative examination, and have signed an informed consent. The lower age limit of 21 years is intended to ensure documentation of refractive stability.
3. Manifest refractive spherical equivalent (MSE) of up to 6.00 diopters (D) at the spectacle plane with refractive cylinder up to 3.00 D.
4. Manifest refraction and LADARWave™ refractions must be within 1.00 D.
5. Best spectacle corrected visual acuity of 20/20 or better in both eyes.
6. Demonstrated refractive stability, confirmed by clinical records. Neither the spherical nor the cylindrical portion of the refraction may have changed more than 0.50D during the 12-month period immediately preceding the baseline examination, as confirmed by clinical records.
7. Soft contact lens users must have removed their lenses at least 2 weeks before baseline measurements. Hard contact lens users (PMMA or rigid gas permeable lenses) must have removed their lenses at least 4 weeks prior to baseline measurements and have 2 central keratometry readings and 2 manifest refractions taken at least 1 week apart that do not differ by more than 0.50 D in either meridian; mires should be regular.
8. Subject must expect to be located in the greater Washington DC area for a 12 month period post-operatively.
9. Consent of the subject's command (active duty) to participate in the study.
10. Access to transportation to meet follow-up requirements

Exclusion Criteria:

1. Female subjects who are pregnant, breast-feeding or intend to become pregnant during the study. Female subjects will be given a urine pregnancy test prior to participating in the study to rule out pregnancy. [Pregnancy and breastfeeding are contraindications to refractive surgery in general, including epi-lasik, whether participating in this study or not]
2. Concurrent topical or systemic medications that may impair healing, including corticosteroids, antimetabolites, isotretinoin (Accutane), amiodarone hydrochloride (Cordarone) and/or sumatripin (Imitrex).
3. Medical condition(s), which, in the judgment of the investigator, may impair healing, including but not limited to: collagen vascular disease, autoimmune disease, immunodeficiency diseases, and ocular herpes zoster or simplex.
4. Active ophthalmic disease, neovascularization of the cornea within 1mm of the intended ablation zone, or clinically significant lens opacity.
5. Evidence of glaucoma or an intraocular pressure greater than 22 mm Hg at baseline.
6. Evidence of keratoconus, corneal irregularity, or abnormal videokeratography in either eye.
7. History of recurrent erosions or epithelial basement dystrophy.
8. Patients with known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course.
9. Any physical or mental impairment that would preclude participation in any of the examinations.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-11; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of Epi-LASIK | 12 months after procedure

CONTACTS AND LOCATIONS:
Overall Officials: KRAIG S. BOWER, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Center for Refractive Surgery, Washington D.C., District of Columbia, United States